CLINICAL TRIAL: NCT03596372
Title: An Open-label, Phase 1, First-in-human, Dose Escalation and Expansion Study to Evaluate the Safety, Tolerability, Pharmacokinetics, Pharmacodynamics and Tumor Response Profile of the Anti-CEACAM6 Antibody BAY1834942 in Patients With Advanced Solid Tumors
Brief Title: Study of BAY1834942 in Patients With Solid Tumors
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Bayer (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Sequential | Masking: None | Purpose: Treatment
Other Study IDs: 18650; 2018-002561-19 (EudraCT Number)
Record Dates: First submitted 2018-06-26; First posted 2018-07-23 (Actual); Last update posted 2022-06-02 (Actual); Status verified 2022-05

CONDITIONS: Advanced CEACAM6-expressing Solid Tumors
Keywords: First-in-human; Immuno-oncology; CEACAM6; Checkpoint inhibition

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (5):
- Patients with Solid tumors (Experimental): Dose escalation with patients having solid tumors. Patients receive escalating doses of BAY1834942 intravenously for 1 hour on Day 1 of each 21-day cycle (Q3W). If the Q3W scheme does not result in sufficient exposure, the scheme is replaced with an once-weekly (QW) dosing scheme.
  Interventions: Drug: BAY1834942
- Patients with Gastric cancer (Experimental): Expansion with patients having gastric and/or gastroesophageal adenocarcinoma:
  Patients receive BAY1834942 intravenously for 1 hour according to dosing scheme decided in escalation part.
  Interventions: Drug: BAY1834942
- Patients with Colorectal cancer (Experimental): Expansion with patients having colorectal cancer:
  Patients receive BAY1834942 intravenously for 1 hour according to dosing scheme decided in escalation part.
  Interventions: Drug: BAY1834942
- Patients with Non-small-cell-lung cancer (Experimental): Expansion with patients having adeno Non-small-cell-lung cancer:
  Patients receive BAY1834942 intravenously for 1 hour according to dosing scheme decided in escalation part.
  Interventions: Drug: BAY1834942
- Low-dose expansion (Experimental): Expansion with patients having the same cancer type (gastric cancer, or colorectal cancer, or non-small-cell lung cancer) and receive BAY1834942 intravenously for 1 hour according to dosing scheme decided in escalation part with a dose lower than the maximum tolerated dose (MTD).
  Interventions: Drug: BAY1834942

INTERVENTIONS:
Drug: BAY1834942 — Dose escalation:
  Sequential dose levels
  .
  Dose expansion (except for low-dose expansion):
  With maximum tolerated dose (MTD) identified in dose escalation part.
  Other Names: Anti-CEACAM6 antibody

SUMMARY:
This is an open-label, Phase 1, first-in-human, dose escalation and expansion study designed to assess the safety, tolerability, pharmacokinetics, pharmacodynamics and tumor response profile of the anti-Carcinoembryonic-antigen-related-cell-adhesion-molecule-6 (CEACAM6) antibody BAY1834942 in patients with advanced solid tumors known to have a prevalence for CEACAM6 expression.

The study consists of dose escalation and a tumor type-specific expansion.

DETAILED DESCRIPTION:
The primary objectives of the study are to evaluate and characterize the tolerability and safety profile of repeated doses of BAY1834942, and to characterize the pharmacokinetics of BAY1834942 after single dose.

Secondary objectives are to evaluate the tumor response profile, pharmacodynamics, pharmacokinetics and immunogenicity after multiple doses of the drug.

ELIGIBILITY:
Inclusion Criteria:

* Male or female patients aged ≥ 18 years
* Patients with histologically confirmed advanced/ metastatic solid tumors: Dose escalation: solid tumor types with a expression of CEACAM6 (gastric/ GEJ cancer, esophageal cancer, NSCLC, CRC, pancreatic cancer, cervical cancer, breast cancer, bladder cancer, head and neck squamous cell cancer, bile duct cancer); Dose expansion: advanced adeno NSCLC, CRC and gastric/ GEJ adenocarcinoma.
* ECOG-PS of 0 to 1.
* Adequate organ function (bone marrow, liver, kidneys).
* Adequate coagulation function.
* Adequate cardiac function

Exclusion Criteria:

* Patients with active symptomatic or untreated brain metastases; possible exceptions for patients with treated asymptomatic central nervous system metastases
* Active autoimmune disease
* History or evidence of active pulmonary fibrosis, organizing pneumonia, or pneumonitis.
* Risk factors for bowel obstruction or bowel perforation
* History of cardiac disease
* Uncontrolled arterial hypertension despite optimal medical management
* Clinically relevant findings in electrocardiogram
* HIV infection
* Active HBV or HCV infection

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Actual)
Dates: Start 2018-06-19 (Actual); Primary Completion 2020-11-16 (Actual); Study Completion 2021-02-22 (Actual)

PRIMARY OUTCOMES:
Incidence of treatment-emergent adverse events | Up to 40 months
Severity of treatment-emergent adverse events | Up to 40 months
  Using the Common Terminology Criteria for Adverse Events (CTCAE) scale
Cmax of BAY1834942 after single dose | 0 (pre-dose), 0.5, 1, 2, 4, 6, 24, 48, 72, 96, 168, 336 and 504 h after drug in Cycle 1 (cycle length is 21 days)
  Maximum plasma concentration of drug after single dose
AUC(0-504) of BAY1834942 after single dose | 0 (pre-dose), 0.5, 1, 2, 4, 6, 24, 48, 72, 96, 168, 336 and 504 h after drug in Cycle 1 (cycle length is 21 days)
  Area under the plasma concentration curve of drug from 0 to 504 hours after single dose

SECONDARY OUTCOMES:
AUC(0-504),md of BAY1834942 after multiple doses | 0 (pre-dose), 0.5, 1, 2, 4, 6, 24, 48, 72, 96, 168, 336 and 504 h in Cycle 3 (cycle length is 21 days)
  Area under the plasma concentration curve of drug from 0 to 504 hours after multiples doses.
Cmax,md of BAY1834942 after multiple doses | 0 (pre-dose), 0.5, 1, 2, 4, 6, 24, 48, 72, 96, 168, 336 and 504 h in Cycle 3 (cycle length is 21 days)
  Maximum plasma concentration of drug after multiples doses
Overall response rate (ORR) | Up to 40 months
  Percentage of patients whose best response to BAY1834942 is either a Complete response or Partial response, both defined according to RECIST criteria
Leukocyte immune phenotyping | Screening; 0 (pre-dose), 24, 168, 336 h after drug on Day 1 of Cycle 1 (cycle length is 21 days); 0 (pre-dose), 24, 168 h after drug on Day 1 of Cycle 2; 0 (pre-dose), 24 h after drug on Day 1 of Cycle 3; 0 h (pre-dose) on Day 1 of Cycles 4, 6 and 8
  Whole blood flow cytometry (FACS) for characterization of blood leukocytes/ lymphocytes with regard to subpopulations, differentiation and activation before and under treatment in all patients
CEACAM6 receptor occupancy | 0 (pre-dose), 24, 168 and 336 h after drug on Day 1 of Cycle 1 (cycle length is 21 days); 0 h (pre-dose) on Day 1 of Cycle 2
  Total and free CEACAM6 expression levels on blood granulocytes and monocytes as assessed by whole blood flow cytometry (FACS) using 2 different fluorescence-labeled anti-CEACAM6 antibodies either competing or not in CEACAM6 binding with BAY1834942 determined before and under treatment in all dose escalation cohorts
Cytokine levels | Screen.; 0 (pre-dose), 4, 24, 168, 336 h after drug on Day 1 of Cycle 1 (cycle length 21 days); 0 (pre-dose), 4, 24, 168 h after drug on Day 1 of Cycle 2; 0 (pre-dose), 4, 24 h after drug on Day 1 of Cycle 3; 0 h (pre-dose) on Day 1 of Cycles 4, 6 and 8
  Total concentration of proinflammatory and immunostimulatory cytokines and of soluble interleukin 2 receptor in serum derived from whole blood taken before and under treatment in all patients
Ex vivo-stimulated cytokine secretion | 0 h (pre-dose) on Day 1 of Cycles 1, 2, 3, 4, 6 and 8 (cycle length is 21 days)
  Total concentration of selected proinflammatory and immunostimulatory cytokines in culture plasma after 24 hour ex-vivo stimulation of whole blood taken before and under treatment in all patients
Concentration of carcinoembryonic antigens (CEA; tumor marker) in serum | 0 h (pre-dose) on Day 1 of Cycles 1, 2, 3, 4, 6 and 8 (cycle length is 21 days)
  Total concentration of CEA in serum derived from whole blood taken before and under treatment in all patients
Concentration of anti-drug antibodies | Day 1 (pre-dose) of Cycles 1, 2, 3, 4, 6 and subsequent odd-numbered cycles (cycle length is 21 days); 1 Day of End of treatment; 1 Day of Safety Follow-up visit
  Concentration in plasma

CONTACTS AND LOCATIONS:
Overall Officials: Bayer Study Director, Study Director — Bayer
Locations (4):
- United States (2):
  - Sarah Cannon Research Institute, Nashville, Tennessee
  - University of Texas MD Anderson Cancer Center, Houston, Texas
- Princess Margaret Hospital-University Health Network, Toronto, Ontario, Canada
- National University Hospital, Singapore, Singapore

REFERENCES:
- [Derived] Siu LL, Hong DS, Docke WD, Tetzner R, Trautwein M, Phelps C, Willuda J, Yu XQ, Nogai H, Johnson M, Goh BC. A Phase I Study of the Anti-CEACAM6 Antibody Tinurilimab (BAY 1834942) in Patients with Advanced Solid Tumors. Target Oncol. 2025 Jul;20(4):637-649. doi: 10.1007/s11523-025-01154-4. Epub 2025 Jun 4. PMID 40465170
- See also: Click here to find results for studies related to Bayer products — http://clinicaltrials.bayer.com/